CLINICAL TRIAL: NCT06338397
Title: Social & Affective Cognition as Determinant of Social Behavior in Alzheimer's Disease & Associated Disorders
Brief Title: Social & Affective Cognition in Alzheimer's Disease & Associated Disorders
Acronym: SOCIALIZE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: France Alzheimer (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023_0455
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Alzheimer's Disease; Frontotemporal Degeneration (Semantic & Behavioral Variants)
Keywords: Emotions; social cognition; social semantics; neuropsychology; frontotemporal dementia
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Social & affective cognition assessment (Experimental)
  Interventions: Other: SCANN

INTERVENTIONS:
Other: SCANN — Administering 11 tests of social & affective cognition to each participant as well as 6 scales to their study-partner, in order to have a detailed profile of social & affective cognitive abilities that we can correlate to an 3DMRI with resting state procedure.

SUMMARY:
Recent studies have shown that individual neuropsychological scores of patients with Alzheimer's disease and Associated Disorders (ADAD) are only poorly correlated to their behavioral difficulties, such as disinhibition, apathy, social decision-making or vulnerability. Recently, social & affective cognitive disorders have been highlighted as potential cause of social behavioral abnormalities. However, no previous studies have assessed the specific relationship between social & affective cognition & social behavior in ADAD. Our pilot study aims to explore the correlations between core and extended social & affective cognitive processes and social behavior as observed during the neuropsychological examination, as well as to explore the common brain regions involved in those domains.

ELIGIBILITY:
Inclusion Criteria:

* Men and women;
* 40 to 85 years of age (included);
* Registered with the French Social Security;
* Have a study partner. The study partner is required to complete several scales. If the subjects or their study partners are not able to drive, their transport fees will be reimbursed by the promotor.
* Fluent in French, able to read and write;

Exclusion Criteria:

* Participants who have contraindications to perform an MRI scan;
* Participants with significant sensory deficits that are not corrected by suitable devices.
* Participants with dementia caused by a non-neurodegenerative disease, including patients with severe cerebrovascular risk factor load, in the judgment of the investigator;
* Participants with other neurodegenerative disease such as Lewy body dementia and Parkinson's disease;
* Participants with other serious neurological disorder such as brain tumor, stroke, epilepsy, hydrocephalus and any condition which contraindicates, in the investigator's judgment, entry to the study;
* Participants with excessive alcohol intake or drug abuse, in the judgment of the investigator;
* Participants who, in the opinion of the investigator, have a risk of non-compliance to the study procedures;

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-02 (Estimated); Primary Completion 2027-05-02 (Estimated); Study Completion 2027-05-02 (Estimated)

PRIMARY OUTCOMES:
Correlation coefficient between the mini Social cognition & Emotional Assessment - mini-SEA - total score and the Social Behavior Observer Checklist - SBOC - score in all participants. | 1day

SECONDARY OUTCOMES:
Correlation coefficients between the mini Social cognition & Emotional Assessment - mini-SEA - sub scores and the neuropsychological assessment (as measured by the Social Behavior Observer Checklist - SBOC - score in all participants. | 1 day
Correlation coefficient between the SBOC score with MRI markers in all participants | 1 day
Correlation coefficient between mini-SEA sub scores & MRI markers in all participants. | 1 day
Correlation coefficients between mini-SEA sub scores with the SOCIAL50, CBI, ZBS, CSDC, SVS scales in each ADAD and controls groups. | 1 day
Correlation coefficients between SCANN sub-scores and the SBOC, SOCIAL50, CBI, ZBS, CSDC, SVS scales in each ADAD and controls groups. | 1 day

IPD SHARING:
Plan to Share IPD: No